CLINICAL TRIAL: NCT07173335
Title: Comparison of In-person and Virtual Delivery of Healthy Lifestyle Focused Care for People With Chronic Musculoskeletal Conditions Living in Rural Areas: a Non-interiority Randomised Trial.
Brief Title: Integrated Healthy Lifestyle and Pain Care for People With Musculoskeletal Conditions Living in Rural Areas.
Acronym: HeLP-R
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Medical Research Future Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/ETH02857; 2031735 (Other Grant/Funding Number: MRFF 2023 Maternal Health and Healthy Lifestyles Grant Opportunity)
Record Dates: First submitted 2025-08-19; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Musculoskeletal Pain; Osteoarthritis; Low Back Pain
Keywords: nutrition; smoking; alcohol; osteoarthritis; low back pain; chronic pain; overweight; obesity; physical activity; lifestyle risk factors; sleep; physiotherapy
MeSH Terms: conditions — Musculoskeletal Pain; Osteoarthritis; Low Back Pain; Smoking; Chronic Pain; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: A parallel group (two arm, 1:1), pragmatic comparative effectiveness, non-inferiority randomised controlled trial.
Who Masked: Outcomes Assessor
Masking Description: All data will be analysed by an independent statistician blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person physiotherapist-led pain and lifestyle care (Active Comparator): Physiotherapist-led integrated healthy lifestyle and pain care delivered in-person with referral to telephone-based health coaching.
  Interventions: Behavioral: In-person physiotherapist led integrated healthy lifestyle and pain care
- Virtual multidisciplinary pain and lifestyle care (Experimental): Multidisciplinary integrated healthy lifestyle and pain care, involving a physiotherapist, dietitian, and psychologist, delivered remotely by virtual care.
  Interventions: Behavioral: Virtual multidisciplinary integrated healthy lifestyle and pain care

INTERVENTIONS:
Behavioral: In-person physiotherapist led integrated healthy lifestyle and pain care — Participants allocated to in-person intervention will be offered:
  A) Up to four in-person physiotherapist consultations (up to one hour in duration) over 12 weeks (weeks 1, 3, 6, and 12);
  B) Tailored pain education and healthy lifestyle education and resource bundles, including video content, web resources and interactive tools sent to participants via email or text;
  C) Referral to telephone-based population wide health behaviour change support services, the NSW Get Healthy Coaching and information service and the Quitline for smokers, by the week 12 consultation (up to 6 telehealth consultations).
  Total = up to 10 consultations over 6 months.
  Arms: In-person physiotherapist-led pain and lifestyle care
Behavioral: Virtual multidisciplinary integrated healthy lifestyle and pain care — Participants allocated to the virtual multidisciplinary intervention will receive:
  A) 10 consultations over 6 months with a multidisciplinary team, including a minimum 4 with a physiotherapist (week 1, 3, 6, 12) and remainder with a dietitian and/or psychologist, tailored to participants needs. Virtual care consultations may be individual or joint multidisciplinary sessions conducted on standard virtual care platforms used by NSW Health. Consultation will be up to one hour in duration, or use an equivalent total duration with a higher frequency schedule. Where appropriate, participants may be referred to alcohol or smoking cessation support, including individualised virtual or telephone-based counselling with access to nicotine replacement therapy;
  B) Tailored pain education and healthy lifestyle education and resource bundles, including video content, web resources and interactive tools sent to participants via email or text.
  Arms: Virtual multidisciplinary pain and lifestyle care

SUMMARY:
This study aims to compare the effects of an in-person physiotherapist-led lifestyle-focused pain care intervention with a virtual multidisciplinary lifestyle-focused pain care intervention on pain impact in people with musculoskeletal conditions and lifestyle risks.

Adults residing in rural and regional locations in New South Wales (AUS) with musculoskeletal conditions (low back, knee or hip pain) recruited from hospital outpatient services (physiotherapy, emergency or orthopaedics) or in response to social media advertisements. Eligible consenting participants will be randomised in a 1:1 ratio to receive either in-person physiotherapy lifestyle intervention or the virtual enabled multidisciplinary intervention. Randomisation will be conducted using an electronic central randomisation service to ensure concealment of treatment allocation.

Participants in both arms (in-person and virtual care) will have up to 10 consultations over six months and follow similar principles based on the previous Healthy Lifestyle for Pain (HeLP) intervention, but differ in their mode of delivery and access to multidisciplinary care.

Participant data will be collected at baseline and weeks 12, 26, 39 and 52. The primary outcome will be Pain Impact measured using the Patient-Reported Outcomes Measurement Information System (PROMIS-29). The secondary outcomes will include participant's health behaviors and mediating outcomes, economic outcomes, process outcomes and adverse events.

DETAILED DESCRIPTION:
One in three Australians experience a musculoskeletal condition, with rural residents experiencing 10% to 30% greater burden. People with musculoskeletal conditions also experience higher rates of chronic health problems and higher prevalence of lifestyle risks (overweight, smoking, physically inactive and poor diet). As many as 75% of people with musculoskeletal conditions have three or more lifestyle risk factors, and those living in rural and remote areas have up to 10% increased prevalence of such risks compared to those living in metropolitan or regional areas. Poorer access to health services for musculoskeletal conditions means patients have higher attendance to emergency departments and increased hospitalisations, which also puts additional strain on tertiary healthcare systems. These factors contribute to a greater burden of musculoskeletal disease in rural populations that is 1.4 times higher than metropolitan populations.

Given the links between musculoskeletal conditions and lifestyle risks, and evidence from meta-analyses, many clinical practice guidelines recommend care for musculoskeletal conditions integrates a focus on lifestyle risks (e.g. weight or smoking). Moreover, surveys of patients with co-existing musculoskeletal conditions and lifestyle risks indicate that most have a preference for integrated care that addresses lifestyle risks. Despite this, less than 25% of such patients receive any support to improve lifestyle. The failure of health services to integrate care for pain and lifestyle risks is a missed opportunity to provide treatment that offers optimal therapeutic benefit for musculoskeletal conditions, supports prevention of chronic diseases, and provides patient-centred care.

A recent trial showed that integrating a healthy lifestyle focus into care for chronic back pain achieved larger improvements in disability, mental health and quality of life, compared to guideline recommended physiotherapy care only (without a lifestyle focus). Participants provided with at least 50% of the lifestyle intervention had large clinically meaningful benefit, suggesting better access to treatment may have large population benefit. Process evaluation of the trial revealed that patients wanted more flexible delivery options to access the intervention, including digital and virtual care options. In response to patient input, about better access to treatment, the HeLP-R trial was designed to compare following two delivery modalities of the program.

* An in-person physiotherapist-led model and referral to a telephone-based health coaching. This intervention aligns with how physiotherapist care is normally delivered in outpatient settings.
* A multidisciplinary model delivered remotely by virtual care, including physiotherapy, dietitian, psychology with additional smoking cessation or alcohol counselling, based on patient health needs. This intervention aligns with feedback from patients and clinicians to provide comprehensive yet flexible care.

MODEL OF CARE:

The model of care being tested across the two delivery modalities includes two core principles to support the integration of healthy lifestyle support into pain care: 1) Learning about pain and its causes; and 2) supporting effective behaviour change for healthy lifestyle.

* 'Learning about pain' is supported in clinical consultations and with education resources. Learning about pain is for clinicians and participants. Clinicians aim to learn about the participant's journey, their pain history and understanding and beliefs about pain. For participants, learning about pain aims to create conceptual change about the causes of pain, provide reassurance about the safety of movement, introduce lifestyle as a potential influence of musculoskeletal pain, and develop motivation to undertake self-management plan focussed on appropriate lifestyle targets. Clinical consultations use principles of motivational interviewing and psychoeducation and are guided by program specific communication aids. Educational resources (electronic and hard copy) are provided to participants in interactive and reflective formats to reinforce learning concepts.
* 'Supporting effective behaviour change' involves co-development of a tailored pain and lifestyle management plan. Clinicians assess the participants stage of change for nominated lifestyle risks (weight, diet, physical activity, smoking, sleep, alcohol) and use behaviour change techniques such as goal setting, action planning, problem solving and monitoring throughout clinical consultations. As appropriate, participants are offered referral to relevant lifestyle risk reduction services which provide telephone-based healthy lifestyle coaching or smoking cessation counselling over 6 calls (each).

ELIGIBILITY:
Inclusion criteria:

* Age 18 years and over, with one or more of the following chronic musculoskeletal conditions (pain or disability due to knee or hip, or non-specific low back pain) present for more than three months;
* Average pain intensity over the last week of 3 or more on a 11-point numerical rating scale OR pain interference of at least 'somewhat' (3 out 5) on item 27 of the PROMIS 29;
* At least one of the following lifestyle risk factors: Body Mass Index of greater than 25kg/m2, less than 30mins of physical activity on five or more days of the week, current smoker or vaper, consumes less than two serves of fruits or five serves of vegetables per day, drinks more than 10 standard drinks in a week, or more than 4 standard drinks on any one day, or 'poor' or 'very poor' sleep quality for item 6 of the Pittsburg Sleep Quality Index.

Exclusion criteria:

* Receiving healthcare for ALL eligible lifestyle risks;
* Had bariatric surgery in the last 12 months or have planned bariatric surgery in the next 6 months;
* Have planned orthopaedic surgery in the next 6 months;
* Cannot actively or safely engage in the intervention or study procedures due to a medical comorbidity or constraint (e.g. impaired cognition, unable to use telehealth services, attend appointments, or adapt meals or activity);
* Pain due to suspected serious cause, (e.g spinal infection, cancers, fracture, systemic rheumatic disease, cauda equina syndrome, diagnosis of radiculopathy);
* Pregnant or planning pregnancy in the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Pain Impact | Baseline (enrolment), week 12, 26, 39 and 52.
  Pain Impact is measured using the Patient-Reported Outcomes Measurement Information System (PROMIS-29). PROMIS-29 is a validated self-report measure that assesses pain, function, and well-being in physical, mental, and social domains. The Pain Impact Score (range 8-50) uses pain intensity, physical function, and pain interference subdomains.

SECONDARY OUTCOMES:
Pain Intensity | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported (PROMIS -29 subdomain); average pain score in the last 7 days on a 0 to 10 numerical rating scale.
Physical Function | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; PROMIS -29 subdomain (4 items measured from 1 to 5 in ability to complete, total score 20).
Depression | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; PROMIS -29 subdomains
Anxiety | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; PROMIS -29 subdomains
Sleep disturbance | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; PROMIS -29 subdomain.
Health-related quality of life | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported, European Quality of Life 5 Dimensions 5 Level Questionnaire
Weight | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported weight (kilograms) to the nearest gram.
Pain self-efficacy | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; Pain Self-Efficacy Questionnaire 2. Two item self-efficacy questionnaire how confident you are that you can do certain activities despite the pain (scale 0-6).
Physical activity levels | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; Global Physical Activity Questionnaire (GPAQ), reported as overall physical activity (MET-mins/week), proportion meeting recommended activity and levels of activity for work, travel and recreation.
Diet quality | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-Reported; Dietary Guidelines Index.
Smoking status | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; adapted from the NSW Health Population Survey smoking status question (including vaping) and Fagerstrom nicotine dependance question.
Alcohol Consumption | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; Alcohol Use Disorders Identification Test-Concise (AUDIT-C scored 0-12). Reported as a continuous use score and the proportion with risky alcohol consumption (≥4 for men and ≥3 for women).
Pain beliefs | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; Pain Beliefs Questionnaire.
Adverse events | Enrolment until end of treatment, and at week 12, 26, 39 and 52.
  Self-reported; "Since the last time we spoke to you have you had any new medical conditions or an exacerbation of another existing condition?"
  Clinical administrative data collected at all participant consultations.
Pain Interference | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; PROMIS -29 subdomain (4 items measured from 1 to 5 for level of interference, total score 20).
Fatigue | Baseline (enrolment), week 12, 26, 39 and 52.
  Description: Self-reported; PROMIS -29 subdomain (4 items measured from 1 to 5 for feelings of fatigue, total score 20).
Participation | Baseline (enrolment), week 12, 26, 39 and 52.
  Description: Self-reported; PROMIS -29 subdomain (4 items measured from 1 to 5 in ability to participate, total score 20).
Cognition | Baseline (enrolment), week 12, 26, 39 and 52.
  Self-reported; PROMIS -29 subdomain (2 items measured from 1 to 5 for level of difficulty, total score 10).

OTHER OUTCOMES:
Fidelity | Enrolment until end of treatment at 26 weeks
  Process outcome: treatment protocol checklist completed using clinical administrative data and summaries of treatment provided.
Perceived importance | Baseline (enrolment), week 12, 26.
  Mediator:
  Self-reported; 3 items (0-10, numerical rating scale) on perceived importance and benefits of healthy lifestyle change.
Patient Reported Experience Measures | Week 12
  Process outcome: Self-reported; 7 or 10 item (group dependant) Patient Reported Experience Measures Outpatient Questionnaire.
Treatment Engagement (consultations) | Enrolment until end of treatment at Week 26.
  Process outcome: Number of consultations attended by a participant and resources provide, detailed in clinical administrative logs, completed by a treating clinicians.
Treatment Engagement (telephone services) | Week 26.
  Process outcome: Self-reported number of calls completed by a participant with telephone support services, if referred.
Work absenteeism and presenteeism | Baseline (enrolment), week 12, 26, 39 and 52.
  Economic outcome: Self-reported; number of days off paid work, and days spent at work with reduced productivity in the last 3 months.
Healthcare utilization | Baseline (enrolment), week 12, 26, 39 and 52.
  Economic outcome: Self-reported; type and number of encounters of health care services and carer support services utilised for back, knee or hip pain, over the last 3 months reported in a participant itemised diary.
Medication use | Baseline (enrolment), week 12, 26, 39 and 52.
  Economic outcome: Self-reported; name and dose of medicines used for back, knee or hip pain, over the last 3 months reported in a participant itemised diary.
Intervention cost | Enrolment until end of treatment at 26 weeks
  Economics outcome: Intervention delivery costs estimated with clinical administrative captured at clinical encounters and patient reported usage of services, and costed with published standardised rates for clinician time, resources and external services.

CONTACTS AND LOCATIONS:
Locations (1):
- University Centre for Rural Health, University of Sydney, Lismore, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data and data dictionaries will be available for sharing beginning 12 months and ending 3 years following the trial's outcomes article publication. Proposals for data should be directed to the Principal Investigator Associate Professor Christopher Williams, and to gain access requestors will need to sign a data access agreement. Investigators proposed use of the data must also be approved by an independent review committee. Study protocols, statistical analyses plans, and primary and secondary analyses data will be publicly available in open access peer reviewed journal articles or on open science framework.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available beginning 12 months and ending 3 years following the trial's outcomes article publication.
Access Criteria: Researchers can request access to the IPD on request, supporting information will be available in open access peer reviewed journal articles or on open science framework.

REFERENCES:
- [Background] Robson E, Kamper SJ, Hall A, Lee H, Davidson S, da Silva PV, Gleadhill C, Williams CM; HeLP Trial Working Group. Effectiveness of a Healthy Lifestyle Program (HeLP) for low back pain: statistical analysis plan for a randomised controlled trial. Trials. 2021 Sep 22;22(1):648. doi: 10.1186/s13063-021-05591-0. PMID 34551809
- [Background] Robson EK, Kamper SJ, Davidson S, Viana da Silva P, Williams A, Hodder RK, Lee H, Hall A, Gleadhill C, Williams CM. Healthy Lifestyle Program (HeLP) for low back pain: protocol for a randomised controlled trial. BMJ Open. 2019 Sep 3;9(9):e029290. doi: 10.1136/bmjopen-2019-029290. PMID 31481555
- [Background] Mudd E, Davidson SRE, Kamper SJ, Viana da Silva P, Gleadhill C, Hodder RK, Haskins R, Donald B, Williams CM; Healthy Lifestyle Program (HeLP) for Chronic Low Back Pain Trial working group. Healthy Lifestyle Care vs Guideline-Based Care for Low Back Pain: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2453807. doi: 10.1001/jamanetworkopen.2024.53807. PMID 39792385